CLINICAL TRIAL: NCT03730623
Title: Cross-sectoral Rehabilitation for Patients With Intermittent Claudication: Effects and Patient Experience - The CIPIC-Rehab Study (Cross-sectoral Intervention for Patients With Intermittent Claudication)
Brief Title: Cross-sectoral Rehabilitation for Patients With Intermittent Claudication
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Maj Siercke Bergstedt, Principal Investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-17004183
Record Dates: First submitted 2018-10-25; First posted 2018-11-05 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Intermittent Claudication
Keywords: Supervised exercise training; community based intervention; Rehabilitation Program; Cross-sectoral intervention; Interdisciplinary; Mixed Methods Research
MeSH Terms: conditions — Intermittent Claudication

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial with118 participants. Randomization to Control group/standard care or Intervention group: 12 week exercise supervised by physiotherapist, Nurse+ dietitian, pedometer and exercise log-book, smoking cessation and text-message follow up. 6 and 12 month follow up. Primary and secondary endpoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): Usual care. Conservative management of IC
- Intervention (Experimental): Supervised exercise
  Interventions: Behavioral: Supervised exercise training

INTERVENTIONS:
Behavioral: Supervised exercise training — Supervised exercise training as a conservative management of intermittent claudication in a community setting based on cardiac rehabilitation program
  Arms: Intervention

SUMMARY:
Exercise training combined with other lifestyle changes are essential elements in conservative management of patients with Intermittent Claudication (IC). IC is essentially caused by atherosclerosis, which reduces blood flow to the legs and leads to cramping leg pain when walking. Patients suffering from IC may have difficulty in exercising and changing lifestyle without systematic intervention despite the risk of morbidity, mortality and hospitalization. Today, rehabilitation programs, including supervised exercise, exist for patients suffering ischemic heart disease but not for patients with IC, despite evidence that exercise therapy is highly beneficial for patients suffering IC.

The overall aim of the present study is to examine the effect of conservative management of patients with IC provided as a three month, cross-sectoral exercise and lifestyle intervention program based on the already established cardiac rehabilitation program. Outcome will be assessed on walking distance and secondly on lifestyle changes and patient reported outcomes.

Implications:

The project will provide evidence for the effect of cross-sectoral collaborative conservative management of patients with IC, using the existing rehabilitation program already offered to patients suffering ischemic heart disease. Moreover, it will elicit knowledge on patient perceptions of conservative management of IC provided as a proactive cross-sectoral intervention and ways to support patients with IC in adhering to conservative management.

DETAILED DESCRIPTION:
Main study:

Randomized Clinical Trial comparing Cross-sectoral Training Intervention for Patients with Intermittent Claudication with standard care.

Patients will be randomized to the intervention or control group using a computer-generated block randomized allocation scheme.

Sample size:

The expected average base line value of maximal walking distance (MWD) has been set to 120 m and the investigators want to detect a 50% improvement (60 m). There is a wide variance in MWD in this patient group, and consequently the standard deviation (SD) is set at 100 m. With a 5% significance level and 80% power, it will thus be necessary to include 88 patients to detect an improvement of 60 m in MWD in the intervention group at 12-months follow-up, compared to the control group. Owing to the previously mentioned risk of comorbidities, combined with an expected loss to follow-up, a drop-out of 25% must be expected, wherefore the investigators plan is to include 118 patients in total (59 in each group).

Baseline data:

The following data will be collected at inclusion, before randomization:

Demography (age, gender, housing, marital status, socioeconomic status, level of education) Height and weight will be combined to report body mass index (BMI) in kg/m^2, waist circumference, blood pressure.

Cardiovascular risk factors, co-morbidity (Charlson Comorbidity Index), current medications, blood samples (biomarkers, cholesterol, HBa1C), based on consultation measurements.

Lifestyle: Measured by self-reported smoking behavior, daily physical activity: minimum 30 min. walking time daylit or other exercise activity, self-reported Diet Registration and alcohol consumption.

Quality of life: Measured using the Vascu-Quality of Life questionnaire (VascuQol).

Depression and anxiety measured with the Hospital Anxiety and Depression Scale (HADS).

Assessment of patients' individual competencies for self-management is measured by using The Patient Activation Measure" (PAM13).

Maximum walking distance (MWD) and pain-free walking distance (PWD) measured using the standardized Treadmill Walking Test, and Visual Analog Score for pain. Follow-up Treadmill Walking Test is performed by a research assistant for whom it is blinded if patients are in intervention or control group.

Control group - standard care. Patients randomized to the control group will initially receive brief advice regarding exercise therapy (walking), smoking cessation, and preventive medical treatment with antiplatelet therapy and statin. Written information about medication, walking exercise, and a logbook for self-reporting of walking behavior is handed out to the IC patients in the outpatient clinic at the Department of Vascular Surgery, Rigshospitalet.

The intervention group will initially receive individual brief advice regarding exercise therapy, smoking cessation advice/course offerings, and preventive medication with antiplatelet therapy and statin in the outpatient clinic at the Department of Vascular Surgery. Patients will receive written standard information and a pedometer and be asked to self-report walking behavior in a logbook.

In the municipality the intervention group will participate in Supervised Exercise Training and education. This entails that patients will actively engage in groups of 8-10 in 24 supervised physical exercise sessions, each lasting one hour with two weekly sessions. Physiotherapists in the training Centre will supervise participants' training. The exercises include varied forms of physical exercise.

The physiotherapists will measure 6 minutes walking test and chair- stand- test prior to and at completion of the intervention and use the results as a part of an individual motivational interview with each patient after completion of the 24 training sessions. Furthermore, participants will be advised in group sessions by the principle investigator, in a 2-hour long session, about the pathophysiology of IC, medications, lifestyle factors, disease management, quality of life and how to cope with the disease. A clinical dietician will advise participants in a 2-hour long session about healthy diet and atherosclerosis. In addition, participants have access to a 2-4 hour long individual consultation with a dietician. After completion of exercise training, participants are offered personalized motivational follow-up text messages. Content, frequency and duration of the text messages are agreed upon individually for the next 8 months and will be reassessed at 3 and 6-months follow-up.

Sub-study. Qualitative Study. Individual brief interview and questionnaire survey supplemented with focus group interviews of patients participating in the intervention group in the randomized clinical study. A protocol for the study will be drawn up in accordance with the "Consolidated Criteria for Reporting Qualitative Research" (COREQ).

An interview guide will be developed prior to interviewing. The investigators expect to explore the following tentative issues: Patient experiences of the training and teaching sessions, factors facilitating or hindering lifestyle changes, how the use of pedometer, logbook and text messages influenced motivation/adherence, patient satisfaction with the intervention and suggestions for future rehabilitation programs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly diagnosed Intermittent Claudication, referred to dept. of vascular surgery and offered conservative management.
* Citizens in the municipalities of the study.
* Able to understand, read and speak Danish.
* Able to perform physical exercise and informed consent to participate in the trial.

Exclusion Criteria:

* Patients that needs vascular surgery.
* Co-morbidity that hinder participation and to perform physical exercise.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2017-12-05 (Actual); Primary Completion 2020-06 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Maximum Walking Distance on a treadmill | 12 months
  Change from Baseline Maximum Walking Distance at 12 months. Detect an improvement of 60 meters in Maximum Walking Distance in the intervention group compared to the control group, using the standardized Treadmill Walking Test.

SECONDARY OUTCOMES:
Pain-free walking distance on a treadmill | 12 months
  Change of Pain-free walking distance (PWD) in meters, measured using the standardized Treadmill Walking Test compared to the control group.
Quality of Life Measurement | 12 months
  Quality of Life questionnaire (VascuQol). Change from Baseline score at 12 months compared to the control group. 6 questions - level of pain, walking capacity and social activity associated with Intermittent claudication.
Depression and anxiety Measurement | 12 months
  Hospital Anxiety and Depression Scale (HADS).Change from Baseline score at 12 months. Score 0-21. Lowest possible score is better.
Self-management Measurement | 12 months
  The Patient Activation Measure (PAM13).Change from Baseline score at 12 months. More or less activation compared to the control group. More activation is better.
smoking cessation Measurement | 12 months
  Change from Baseline score at 12 months.Smoking cessation or not.
Daily physical activity Measurement | 12 months
  Change from Baseline score at 12 months. More or less active. Minimum 30 min. walking daily.
Diet Registration Measurement | 12 months
  Change from Baseline score at 12 months. More or less healthy diet. Healthy diet score change to a higher percentage where 75% is healthy diet.

CONTACTS AND LOCATIONS:
Overall Officials: Selina Kikkenborg Berg, Professor, Study Director — University of Copenhagen
Locations (1):
- Dept. of Vascular Surgery, Rigshospitalet, University of Copenhagen., Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Siercke M, Jorgensen LP, Missel M, Thygesen LC, Blach PP, Sillesen H, Berg SK. Cross-sectoral rehabilitation intervention for patients with intermittent claudication versus usual care for patients in non-operative management - the CIPIC Rehab Study: study protocol for a randomised controlled trial. Trials. 2020 Jan 21;21(1):105. doi: 10.1186/s13063-019-4032-x. PMID 31964402